CLINICAL TRIAL: NCT00455143
Title: Cognitive Protection - Dexmedetomidine and Cognitive Reserve
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Pilot study initiated to provide support data for main grant GCO 06-0217 funded. only baseline characteristic data collected. no results for this study.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 06-0453
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Delirium; PD; Postoperative Cognitive Dysfunction; POCD
Keywords: Postoperative delirium; PD; Postoperative cognitive dysfunction; POCD
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively. Patients will receive dexmedetomidine until discharge from the PACU.
  Interventions: Drug: Precedex (Dexmedetomidine)
- Placebo (Placebo Comparator): Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively or until discharge from the PACU.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Precedex (Dexmedetomidine) — Dexmedetomidine started prior to surgery and continued for 24 hours postoperatively. Patients will receive dexmedetomidine until discharge from the PACU.
  Other Names: Precedex; Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Placebo — Matching placebo given prior to surgery and continued for 24 hours postoperatively
  Arms: Placebo

SUMMARY:
This is a pilot study to evaluate the effect of dexmedetomidine in the prevention of delirium in non-cardiac surgical patients. The preliminary data regarding the effect of dexmedetomidine on delirium comes from a study underway at Stanford. We propose to randomize fifty patients into two different protocols, one using dexmedetomidine until PACU discharge (hip replacement) and the other using dexmedetomidine for 24 hours in a monitored setting.

DETAILED DESCRIPTION:
Elderly patients who undergo anesthesia and non-cardiac surgery are subject to deterioration of brain function including the development of postoperative delirium (PD) and postoperative cognitive dysfunction (POCD). These disorders cause disability, distress for both patients and their families, are associated with other medical complications and account for significant additional health care costs. We currently use relatively primitive approaches to preventing and treating PD and POCD. The proposed is a pilot study for an NIH grant which was recently submitted. This is a randomized controlled trial of perioperative dexmedetomidine to prevent PD and, potentially, POCD. Fifty patients will be enrolled at Mount Sinai with two different surgeries, either hip replacement or vascular bypass. The patients undergoing hip replacement will receive dexmedetomidine until discharge from the PACU. Vascular surgery patients who are transferred from the PACU to a monitored step-sown unit will continue dexmedetomidine for 24 hours.Participants will be screened for Mild Cognitive Impairment (MCI), and undergo preoperative cognitive testing. Unlike the parent trial, we will test for but will not select for patients with MCI. Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively. Follow up studies will include surveillance for delirium while in the hospital and cognitive testing at 3 months following surgery.

Dexmedetomidine is a drug used for sedation in critically ill patients that provides some pain relief and controls the bodies response to stress. The sedation produced by dexmedetomidine appears more similar to natural sleep than any other drug used for anesthesia and postoperative sedation. Data suggesting that dexmedetomidine can prevent delirium following cardiac surgery and the developing understanding of the causes of PD and POCD suggest that dexmedetomidine will be particularly effective.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years and older
* elective major hip replacement or peripheral vascular (major surgery is defined by a planned 2 day hospitalization)
* ASA physical status I-III
* capable and willing to consent

Exclusion Criteria:

* Cardiac surgery
* Intracranial Surgery
* Emergency Surgery
* Patients with severe visual or auditory disorder/handicaps
* Illiteracy
* Patients with clinically significant Parkinson's Disease
* Patients not expected to be able to complete the 3 month postoperative test
* Sick sinus syndrome without pacemaker
* Hypersensitivity to drug or class
* Current 2nd or 3rd degree AV block
* History of clinically significant bradycardia
* Contraindication to the use of an 2A-agonist
* Presence of a major psychiatric condition such as bipolar disorder, major depression, schizophrenia, or dementia
* ASA physical status IV or V

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Silverstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from September 2006 to March 2008
Groups:
- All Participants: All participants enrolled in study. Information not available per arm. Study never unblinded.
Period: Overall Study
Arm/Group | All Participants
Started | 27
Completed | 21
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Staff was not avail to follow patient | 2
Not completed — No longer met Inclusion Criteria | 1
Not completed — Surgical time, staff not available | 1

BASELINE CHARACTERISTICS:
Population: Missing information for 1 participants
Groups:
- All Participants: All participants enrolled in study. Study never unblinded. Information not available by arms.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Functional Recovery
Time Frame: 3 months post surgery
Population: Main protocol became funded, study terminated, data not collected.
Groups:
- Dexmedetomidine: Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively. Patients will receive dexmedetomidine until discharge from the PACU.
  Precedex (Dexmedetomidine): Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively. Patients will receive dexmedetomidine until discharge from the PACU.
- Placebo: Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively or until discharge from the PACU.
  Precedex (Dexmedetomidine): Participants will be randomized to either dexmedetomidine or placebo which will be started prior to surgery and continued for 24 hours postoperatively. Patients will receive dexmedetomidine until discharge from the PACU.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Functional Recovery
Time Frame: 6 months post surgery
Population: This study terminated because main study became funded, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cognitive Testing
Time Frame: prior to surgery
Population: This study terminated because main study became funded, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cognitive Testing
Time Frame: 3 months post surgery
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cognitive Testing
Time Frame: 6 months post surgery
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Delirium Assessments
Time Frame: prior to surgery
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Delirium Assessments
Time Frame: duration of PACU stay, up to 4 days post-op
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Delirium Assessments
Time Frame: 3 months post surgery
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Delirium Assessments
Time Frame: 6 months post surgery
Population: Main protocol became funded, study terminated, data not collected.
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- All Participants: All participants enrolled in study, data missing for 3 participants. Information not available per arm. Study never unblinded.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 6/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=24)
Hypotension (Cardiac disorders) | 1
Hypoxia (General disorders) | 1
Post-operative Confusion (General disorders) | 1
Cellulitis (Infections and infestations) | 2
Anemia (Blood and lymphatic system disorders) | 3

LIMITATIONS AND CAVEATS:
Investigator passed away. Study team no longer at institution. Study material not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes